CLINICAL TRIAL: NCT04728503
Title: Brief Video-Based Mindful Movement Intervention Prior to Pelvic Exams
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Tracy Greer, Associate Professor, Department of Psychiatry, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: STU-2019-1782
Record Dates: First submitted 2021-01-11; First posted 2021-01-28 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Anxiety State; Pain; Depression
MeSH Terms: conditions — Anxiety Disorders; Pain; Depression

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 5-Minute Mindful Movement Video (Experimental): 5 minute mindful movement video watched in the exam room on an iPad
  Interventions: Behavioral: 5-Minute Mindful Movement Video
- Written Educative Materials (Placebo Comparator): 1 page printed written educative material about mindfulness benefits read for 5 minutes in the exam room
  Interventions: Behavioral: Written Educative Materials

INTERVENTIONS:
Behavioral: 5-Minute Mindful Movement Video — 5 minute video includes a brief verbal introduction to mindfulness and then guides participants through a mindful movement exercise to facilitate grounding in the present moment and activation of the parasympathetic nervous system.
  Arms: 5-Minute Mindful Movement Video
Behavioral: Written Educative Materials — 1 page written educative material about the benefits of mindfulness to serve as a control.
  Arms: Written Educative Materials

SUMMARY:
This study endeavors to implement a brief video-based mindfulness intervention within a clinic setting for women undergoing pelvic examinations, in hopes of reducing state anxiety and pain intensity during pelvic exams and improving overall exam satisfaction and likelihood to return for follow-up exams. This will be a pilot study will take place the University of Texas Southwestern (UTSW) Lowe Foundation Center for Women's Preventative Health Care. There will be a treatment and a control arm, estimated 50 women per group.

DETAILED DESCRIPTION:
Participants will be randomly assigned to either a treatment group or a control group. Treatment group will receive a 5-minute mindful movement video-based intervention before their previously scheduled pelvic exam. Control group will not receive the mindful movement video-based intervention and will instead be given a handout about the benefits of mindfulness to read prior to the pelvic exam. Control group will be given access to the mindfulness intervention via an online link upon completion of participation in the study to ensure they are provided the opportunity to benefit from mindfulness practice.

Participants will be recruited from a group of female patients at the Lowe Foundation Center who have already been scheduled for an upcoming pelvic exam. Therefore the pelvic exam procedure itself is standard of care, the experimental piece is the mindfulness intervention before the pelvic exam - either the video, or the written educational materials depending on whether participants are randomly assigned to the treatment or control group.

ELIGIBILITY:
Inclusion Criteria:

1. Female
2. Age of 18+ years
3. Scheduled physical evaluation including pelvic exam at UT Southwestern's Lowe Foundation Center for Women's Preventative Health Care.

Exclusion Criteria:

1. Participants who are unable to read, speak, write or understand verbally spoken English
2. Participants who are blind or otherwise visually impaired will be excluded due to nature of video intervention.
3. Participants who are pregnant will be excluded from the study.
4. Individuals presenting to the clinic for an acute pain reason will be excluded from the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2020-12-08 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Visual Analogue Scale - Anxiety 1 (Change in Anxiety) | baseline, pre-intervention/procedure
  Using an iPad, participant slides a bar on a scale to the right or left to indicate level of anxiety. All the way to the right indicates highest anxiety (100) all the way to the left indicates no anxiety (0). Higher number indicates worse outcome/more anxiety.
Visual Analogue Scale - Anxiety 2 (Change in Anxiety) | immediately after the intervention
  Using an iPad, participant slides a bar on a scale to the right or left to indicate level of anxiety. All the way to the right indicates highest anxiety (100) all the way to the left indicates no anxiety (0). Higher number indicates worse outcome/more anxiety.
Visual Analogue Scale - Anxiety 3 (Change in Anxiety) | immediately after the procedure
  Using an iPad, participant slides a bar on a scale to the right or left to indicate level of anxiety. All the way to the right indicates highest anxiety (100) all the way to the left indicates no anxiety (0). Higher number indicates worse outcome/more anxiety.
Visual Analogue Scale - Pain 1 | baseline, pre-intervention
  Using an iPad, participant slides a bar on a scale to the right or left to indicate level of pain. All the way to the right indicates highest pain (100) all the way to the left indicates no pain (0). Higher number indicates worse outcome/more pain.
Visual Analogue Scale - Pain 2 | immediately after the procedure
  Using an iPad, participant slides a bar on a scale to the right or left to indicate level of pain. All the way to the right indicates highest pain (100) all the way to the left indicates no pain (0). Higher number indicates worse outcome/more pain.

SECONDARY OUTCOMES:
Patient Health Questionnaire (PHQ-9) | baseline, pre-intervention/procedure
  Depression symptom severity scale; 9 items with a total score ranging from 0-27, higher score means a greater number of depressive symptoms endorsed. Scores of 5, 10, 15, and 20 represent cutpoints for mild, moderate, moderately severe and severe depression, respectively.
Exam Satisfaction Survey | immediately after the procedure
  Assess overall patient satisfaction with exam, and likelihood to attend future appointments
Mindfulness Perceptions Survey | immediately after the procedure
  Treatment group completes a survey regarding perceptions of mindfulness video
Physician Experience Survey | immediately after the procedure
  Physician who completes the pelvic exam will rate their experience completing the pelvic exam

CONTACTS AND LOCATIONS:
Overall Officials: Tracy Greer, PhD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No
We do not have a formal data sharing plan; however, if investigators are interested in using these data, they may contact us to determine if that may be possible.